CLINICAL TRIAL: NCT04336891
Title: Pilot Retrospective Study on the Effect of Testosterone Treatment on Clitoral Arteries' Hemodynamic Parameters.
Brief Title: Effect of Testosterone Treatment on Clitoral Arteries' Hemodynamic Parameters.
Acronym: TESTOFSD
Status: Completed | Type: Observational
Sponsor: University of Florence (Other)
Responsible Party: Principal Investigator, Linda Vignozzi, MD, Associate Professor of Endocrinology; Chief of Andrology, Women's Endocrinology and Gender Incongruence, Careggi Hospital, University of Florence
Other Study IDs: FEMENDO1; 14457_oss (Other: AOU Careggi Ethics Committee)
Record Dates: First submitted 2020-04-03; First posted 2020-04-07 (Actual); Last update posted 2020-04-07 (Actual); Status verified 2020-04

CONDITIONS: Hypoactive Sexual Desire Disorder; Vulvovaginal Disease; Menopause Related Conditions; Dyspareunia (Female Excluding Psychogenic); Hypoestrogenism; Arousal Disorders, Sexual
Keywords: testosterone; female sexual dysfunction; genital vascularization; clitoris; dyspareunia
MeSH Terms: conditions — Sexual Dysfunctions, Psychological; Dyspareunia | interventions — Estradiol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Hypoactive Sexual Desire Disorder: Women with Hypoactive Sexual Desire Disorder (HSDD, n=23)
  Interventions: Drug: Testosterone gel
- Moderate to severe VVA: Women with dyspareunia due to moderate to severe vulvovaginal atrophy (VVA) (n=12)
  Interventions: Drug: Estradiol ovules
- Mild to moderate VVA: Women with dyspareunia due to mild to moderate VVA (n=37)
  Interventions: Drug: Moisturizer
- HSDD + VVA: Women with HSDD reporting also significant dyspareunia due to moderate to severe VVA (n=9).
  Interventions: Drug: Testosterone gel + Estradiol ovules

INTERVENTIONS:
Drug: Testosterone gel — Transdermal 2% T gel applied once daily to the thighs or lower abdominal/pubic area (300 mcg T per day) for 6 months
  Groups: Hypoactive Sexual Desire Disorder
Drug: Estradiol ovules — Intravaginal estradiol ovules taken daily for 2 weeks and afterwards twice a week, for 6 months
  Groups: Moderate to severe VVA
Drug: Moisturizer — Local non-hormonal moisturizers applied regularly every 2-3 days and lubricants as needed
  Groups: Mild to moderate VVA
Drug: Testosterone gel + Estradiol ovules — Transdermal 2% T gel applied once daily to the thighs or lower abdominal/pubic area (300 mcg T per day), plus Intravaginal estradiol ovules taken daily for 2 weeks and afterwards twice a week, for 6 months
  Other Names: Estradiol
  Groups: HSDD + VVA

SUMMARY:
The regulation of clitoral vascularization by sex steroids is still under-investigated. We aimed to explore the effects of 6 months transdermal Testosterone (T) therapy on clitoral color Doppler ultrasound (CDU) parameters in pre- and postmenopausal women with female sexual dysfunction (FSD). In order to do that, we retrospectively recruited n=81 women with FSD, divided into 4 groups according to different treatments followed as per clinical practice, for 6 months: transdermal systemic 2% T gel; local estradiol ovules; local non-hormonal moisturizers; transdermal T plus local estrogens.

Our main hypothesis is that systemic T treatment is able to positively modulate clitoral blood flow in basal conditions, specifically to increase clitoral artery Peak systolic velocity (PSV).

DETAILED DESCRIPTION:
Strong clinical evidence supports the use of transdermal systemic testosterone (T) treatment for Hypoactive Sexual Desire Disorder (HSDD) in menopausal women. According to preclinical studies, T is necessary to maintain the functional machinery underlying clitoral arousal response. In hypogonadal men with erectile dysfunction, T replacement therapy is able to improve penile vasodilation as assessed by using color Doppler ultrasound (CDU). On the other hand, the regulation of clitoral vascularization by sex steroids is still under-investigated.

We aimed to explore the effects of 6 months T therapy on clitoral CDU parameters and sexual function in pre- and postmenopausal women with female sexual dysfunction (FSD).

Adult heterosexual women attending our clinic for sexual concerns were retrospectively recruited. A subgroup of sexually active patients with FSD (n=81) was divided into 4 different groups according to different treatments followed as per clinical practice: women with Hypoactive Sexual Desire Disorder (HSDD) treated with off-label transdermal 2% T gel once daily (300 mcg T per day, n=23); women with dyspareunia due to moderate to severe vulvovaginal atrophy (VVA), treated with local estrogens (estradiol ovules) taken daily for 2 weeks and afterwards twice a week (n=12); women with dyspareunia due to mild to moderate VVA, treated with non-hormonal moisturizers every 2-3 days (n=37); women with HSDD reporting also significant dyspareunia due to moderate to severe VVA, treated with combined therapy (transdermal T and local estrogens) (n=9). Patients underwent physical, laboratory, uterine and genital (clitoral and uterine arteries) CDU examinations, and completed the Female Sexual Function Index (FSFI). at baseline and after 6 months.

Our main hypothesis is that systemic T treatment is able to positively modulate clitoral blood flow in basal conditions, specifically to increase clitoral artery Peak systolic velocity (PSV).

ELIGIBILITY:
Inclusion Criteria:

* being heterosexual.

Exclusion Criteria:

* history of drug or alcohol abuse
* a diagnosis of uncontrolled or unstable mental or organic disease.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Pre- and postmenopausal women who attended our outpatient clinic at Andrology, Women's Endocrinology and Gender Incongruence Unit, University of Florence (Florence, Italy) for sexual concerns.
Sampling Method: Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2019-03-20 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Changes of clitoral artery peak systolic velocity (PSV) in women treated with testosterone gel | 6 months
  parameter evaluated at clitoral color Doppler ultrasound
Changes of clitoral artery pulsatility index (PI) in women treated with testosterone gel | 6 months
  parameter evaluated at clitoral color Doppler ultrasound
Changes of clitoral artery acceleration (ACC) in women treated with testosterone gel | 6 months
  parameter evaluated at clitoral color Doppler ultrasound

SECONDARY OUTCOMES:
Difference in changes of clitoral artery PSV among the 4 intervention groups | 6 months
Difference in changes of clitoral artery PI among the 4 intervention groups | 6 months
Difference in changes of clitoral artery ACC among the 4 intervention groups | 6 months

OTHER OUTCOMES:
Changes in Female Sexual Function Index (FSFI) Total, desire, arousal, lubrication, orgasm, satisfaction and pain scores, in women treated with transdermal Testosterone | 6 months
Changes in serum total Testosterone levels in women treated with transdermal Testosterone | 6 months
  Women were asked to have blood samples drawn in the morning, after an overnight fast, during the early follicular phase (if premenopausal)
Changes in serum total Sex Hormone Binding Globulin (SHBG) levels in women treated with transdermal Testosterone | 6 months
  Women were asked to have blood samples drawn in the morning, after an overnight fast, during the early follicular phase (if premenopausal)
Difference in changes of - Total cholesterol, high-density lipoprotein cholesterol, triglycerides, glycated hemoglobin, fasting glucose and insulin levels among the 4 intervention groups | 6 months
  Women were asked to have blood samples drawn in the morning, after an overnight fast

CONTACTS AND LOCATIONS:
Locations (1):
- Andrology, Women's Endocrinology and Gender Incongruence Unit, University of Florence, Azienda Ospedaliero-Universitaria Careggi, Florence, Italy

REFERENCES:
- [Background] Scavello I, Maseroli E, Di Stasi V, Cipriani S, Verde N, Magini A, Maggi M, Vignozzi L. Nomegestrol acetate/17beta-estradiol does not negatively alter the vascular resistance of clitoral arteries: a prospective, exploratory study. Int J Impot Res. 2020 Mar;32(2):239-247. doi: 10.1038/s41443-019-0162-7. Epub 2019 Jul 1. PMID 31263248
- [Background] Maseroli E, Scavello I, Vignozzi L. Cardiometabolic Risk and Female Sexuality-Part II. Understanding (and Overcoming) Gender Differences: The Key Role of an Adequate Methodological Approach. Sex Med Rev. 2018 Oct;6(4):525-534. doi: 10.1016/j.sxmr.2018.03.004. Epub 2018 Apr 13. PMID 29661689
- [Background] Davis SR, Baber R, Panay N, Bitzer J, Perez SC, Islam RM, Kaunitz AM, Kingsberg SA, Lambrinoudaki I, Liu J, Parish SJ, Pinkerton J, Rymer J, Simon JA, Vignozzi L, Wierman ME. Global Consensus Position Statement on the Use of Testosterone Therapy for Women. J Clin Endocrinol Metab. 2019 Oct 1;104(10):4660-4666. doi: 10.1210/jc.2019-01603. PMID 31498871
- [Derived] Cipriani S, Maseroli E, Di Stasi V, Scavello I, Todisco T, Rastrelli G, Fambrini M, Sorbi F, Petraglia F, Jannini EA, Maggi M, Vignozzi L. Effects of testosterone treatment on clitoral haemodynamics in women with sexual dysfunction. J Endocrinol Invest. 2021 Dec;44(12):2765-2776. doi: 10.1007/s40618-021-01598-1. Epub 2021 Jun 12. PMID 34118018